CLINICAL TRIAL: NCT03786003
Title: Lobectomy for Clincial Stage T1N0M0 Solid NSCLC by VATS Versus Thoracotomy
Brief Title: ELobectomy for NSCLC by VATS Versus Thoracotomy (ECTOP-1007)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNVT
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Video-Assisted Thoracic Surgery; Thoracotomy; Early-stage NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thoracic Surgery, Video-Assisted; Thoracotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VATS (Experimental): Video-assisted thoracoscopic surgery
  Interventions: Procedure: VATS
- Thoracotomy (Active Comparator): Open surgery
  Interventions: Procedure: Thoracotomy

INTERVENTIONS:
Procedure: VATS — Standard video assisted thoracic surgery, no use of rib-spreader.
  Arms: VATS
Procedure: Thoracotomy — Standard thoracotomy
  Arms: Thoracotomy

SUMMARY:
This study is one of Eastern Cooperative Thoracic Oncology Projects (ECTOP-1007). The goal of this study is to determine video-assisted thoracoscopic surgery is non-inferior to thoracotomy in terms of disease-free survival for solid clinical stage T1N0M0 NSCLC.

DETAILED DESCRIPTION:
It is a randomized clinical trial comparing video-assisted thoracoscopic surgery (VATS) with thoracotomy for solid clinical stage T1N0M0 NSCLC. The primary objective of the study is to determine that VATS is non-inferior to thoracotomy in terms of disease-free survival (DFS). Secondary objectives are to compare VATS and thoracotomy for overall survival (OS), perioperative complications, pain levels and quality of life.

Although there are numerous retrospective studies have indicated feasibility and effectiveness of VATS, no data has been reported from those prospective and randomized clinical trials with prognostic indicators as the primary objective. Whether VATS is non-inferior to thoracotomy in terms of survival is still unclear. Therefore, we design this trial by recruiting patients in clinical stage T1N0M0 with solid mass on computed tomography (CT). To determine the clinical stage, CT scans will be performed routinely and PET-CT/EBUS-TBNA/mediastinoscopy will be conducted in patients with suspected positive mediastinum lymph node or distant metastases. Detailed inclusion criteria include clinical stage T1N0M0 and surgical resectable, solid appearance on CT, age 18 to 75 year and signed informed consent. Exclusion criteria includes not NSCLC in pathologic analysis, no lobectomy or sublobar resection, history of other malignant tumors within 5 years, history of thoracic surgery or unsuitable for VATS and previous radiation or chemotherapy.

In our previous data, the 3-year DFS for cT1N0M0 patients with solid mass who were subjected to thoracotomy (lobectomy or sublobar resection) was 77.9%. If the 3-year DFS of VATS arm is not less than 70.9%, the VATS arm will be regarded to be non-inferior to thoracotomy. A sample size of at least 1086 participants is required for performance equal to 80%, α-level equal to 0.025, 1:1 recruitment and considering a dropout rate of 10%. Participants will be randomly assigned to either group using a random table.

Lobectomy or sublobar resection will be conducted by standard procedures at the discretion of the surgeon. Each participating surgeon will be evaluated by the trial committee to ensure proper surgical technique. If the VATS is diverted to thoracotomy intraoperartively, the reason will be recorded, and the cause will still be analyzed in an intention-to-treat analysis. Patients will be follow-up every 6 months to 3 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage T1N0M0 and surgical resectable.
* Solid appearance on computed tomography scan.
* Age 18 to 75 year.
* Signed the informed consent form.

Exclusion Criteria:

* Not NSCLC in pathological analysis.
* Not lobectomy or sublobar resection.
* History of other malignant tumors within 5 years.
* History of thoracic surgery or unsuitable for VATS.
* Previous radiation or chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1086 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2025-02-09 (Estimated); Study Completion 2028-02-09 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years after the surgery
  Disease-free survival means the period after surgery when no disease can be detected.

SECONDARY OUTCOMES:
Overall survival | 3 years after the surgery
  Overall survival means the period after surgery when a patient doesn't die directly from lung cancer or an unrelated cause.
Rate of patients with perioperative complication | 1 month after surgery
  The perioperative complication includes wound infection, hemorrhage, infection, pleural effusion, pneumothorax, cardiovascular problem and etc within a month after surgery.
Pain degree and quality of life | 1 years after the surgery
  Numerical rating score (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Shanghai Cancer Center Chen, Ph.D, Principal Investigator — Shanghai Cancer Center
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Inform Consent Form, Clinical Study Report would be shared every 3 months after the study begin.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Every 3 months after the study begin.